CLINICAL TRIAL: NCT06776042
Title: Upper Airway Inflammation and Olfaction: Mechanisms of Loss and Recovery
Acronym: IMMUNODOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/15DEC/484
Record Dates: First submitted 2024-12-06; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic rhinosinusitis patients (Experimental): Patients suffering from chronic rhinosinusitis will undergo smell testing as well as nasal brushing of the olfactory cleft
  Interventions: Other: Nasal brushing of the olfactory cleft; Other: Smell testing

INTERVENTIONS:
Other: Nasal brushing of the olfactory cleft — Nasal brushing of the olfactory cleft
Other: Smell testing — Smell testing using the Sniffin' Sticks Test

SUMMARY:
The goal of this clinical trial is to understand the mechanisms leading to olfactory dysfunction (OD) in chronic rhinosinusitis (CRS). The main questions it aims to answer are:

* Is the type 2 inflammation impacting the olfactory epithelium regeneration, leading to OD?
* Does a treatment interfering with one of the major T2 inflammatory cytokines, have an impact on the mechanisms of OD in CRS?

Participants will undergo olfactory testing and nasal brushing before and after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least two of the following symptoms: nasal obstruction, rhinorrhoea, smell loss, facial pain for 12 weeks.
* Endoscopic visualisation of bilateral sinonasal polyps
* SSI (TDI) < 30.75 and decreased sense of smell subjectively
* Eosinophilia > 300/μl of blood Ku/l
* On a stable nasal steroid treatment for at least 4 weeks

Exclusion Criteria:

* Active smoking
* Primary and secondary immune deficiencies
* Ciliary diseases (cystic fibrosis, primary ciliary diskinesia)
* History of or current nasal malignancies
* < 18 years and > 70 years
* Patients unable to express consent
* Use of systemic corticosteroids for < 4 weeks before visit 1 • Use of systemic or local antibiotics for < 4 weeks before visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Genetic profile comparison after single-cell RNA sequencing | Through study completion, an average of 2 years
  The primary objective of this study is to compare the genetic profile of the olfactory epithelium from T2 CRSwNP patients harvested with a nasal brush, to the olfactory epithelium from healthy controls (HC) by means of RNA sequencing.

SECONDARY OUTCOMES:
Functional characterization of olfactory epithelium | Through study completion, an average of 2 years
  The secondary objectives are to characterize the OE of T2 CRSwNP patients in a functional way by means of immunocytochemistry (ICC), calcium imaging, and proliferation assays, and to compare the results with healthy controls, patients with non-inflammatory OD and non-T2 CRSsNP.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Hox, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium